CLINICAL TRIAL: NCT06229158
Title: Assessment of the Quality and Sexual Health Needs of Patients with Advanced-stage Cancer
Acronym: INTIMI-K
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0695
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Advanced Cancer; Sexual Satisfaction
Keywords: sexual health; palliative cancer patients; identification of needs
MeSH Terms: conditions — Orgasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients' group: Patients diagnosed with advanced solid or hematological cancers, whether or not undergoing specific treatment for the ongoing oncological condition and having a cancer diagnosis for more than 3 months (baseline diagnosis consultation).
  Interventions: Other: Sexual satisfaction questionnaire for patients
- Partners' of life group: Partners' of life group of patients' diagnosed with advanced solid or hematological cancers, whether or not undergoing specific treatment for the ongoing oncological condition and having a cancer diagnosis for more than 3 months (baseline diagnosis consultation).
  Interventions: Other: Sexual satisfaction questionnaire for patients' life partner

INTERVENTIONS:
Other: Sexual satisfaction questionnaire for patients — Completion by patients of a 28-item ad-hoc questionnaire evaluating their sexual satisfaction, alone or with the help of one of the researchers.
  Each item is rated using a Likert-type scale from 1 to 5. The maximum score is 140, the minimum score is 28. A low score reflects a good level of sexual satisfaction.
  Participants who have agreed to take part in the qualitative part of the study will be contacted within a few days of inclusion to arrange an appointment for a semi-structured individual interview.
  Groups: Patients' group
Other: Sexual satisfaction questionnaire for patients' life partner — Completion by the patients' life partner of a 30-item ad-hoc questionnaire evaluating their sexual satisfaction, alone or with the help of one of the researchers.
  Each item is rated using a Likert-type scale from 1 to 5. The maximum score is 140, the minimum score is 28. A low score reflects a good level of sexual satisfaction.
  Participants who have agreed to take part in the qualitative part of the study will be contacted within a few days of inclusion to arrange an appointment for a semi-structured individual interview.
  Groups: Partners' of life group

SUMMARY:
Sexual health is an important determinant of the overall health of a population, as addressed in the French National Strategy 2017-2030. For a long time neglected in oncology, sexual health is now part of clinical assessments in cancer support care and is fully integrated into practice recommendations. However, existing evidences, though limited, are still suggesting unmet needs during the palliative phase of the disease.

Current literature focuses on the assessment and management of potential issues related to genital cancers - primarily gynecological, breast, and prostate cancers - but also on post-cancer experiences. The sexual health needs of patients in palliative care are understudied, except one study that reports how patients are considering sexuality as an important aspect of their lives, even during the last weeks to days of life.

In the aim of developing an efficient complex intervention for the population of patients with cancer in palliative situations, it is necessary to identify the needs, facilitators, and modalities required for promoting sexual health in this population (beyond the extensively studied cases of genital cancers). A solely patient-centred approach would be limiting, and this objective requires an approach dedicated to the life partners as well.

To assess satisfaction related to sexual health and gain insights regarding the expectations of patients and their partners towards the healthcare system, the study INTIMI-K will utilize a mixed methodology involving the use of a questionnaire, including validated scales, and semi-structured interviews. Patients aged 18 and older, diagnosed with advanced solid or hematological cancers, along with their life partner will be included.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Individuals aged 18 and older,
* Patients diagnosed with advanced solid or hematological cancers,
* Whether or not undergoing specific treatment for the ongoing oncological condition,
* Having a cancer diagnosis for more than 3 months (baseline diagnosis consultation),
* Capable of understanding study-related documents,
* Capable of completing questionnaires,
* Fluent in French,
* Individuals who have not objected to participating in the study.

For partners:

* Individuals aged 18 and older,
* Individuals whose life partner has been diagnosed with advanced solid or hematological cancer for more than 3 months, whether or not they have received treatment,
* Capable of understanding study-related documents,
* Capable of completing questionnaires,
* Fluent in French,
* Individuals who have not objected to participating in the study.

Exclusion Criteria:

* Individuals unable to complete the entire questionnaire due to their clinical condition.
* Individuals under guardians, curators, or legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with advanced solid or hematological cancers, whether or not undergoing specific treatment for the ongoing oncological condition and having a cancer diagnosis for more than 3 months (baseline diagnosis consultation) and their partner of life.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Sexual Health satisfaction assessment | Day 1
  Average scores for the various questions from the different developed ad-hoc questionnaire to assess satisfaction related to sexual health

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre hospitalier de la Croix Rousse, Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Edouard Herriot, Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No